CLINICAL TRIAL: NCT05421845
Title: Prevention of Gestational Diabetes Mellitus With Mobile- and Hospital-based Lifestyle Intervention Among Women of Advanced Maternal Age: a Randomized Controlled Study.
Brief Title: Prevention of Gestational Diabetes Mellitus With Lifestyle Intervention Among Women of Advanced Maternal Age.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BMU2022MX022
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: advanced maternal age; gestational diabetes mellitus; lifestyle intervention; randomized controlled study
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention group (Experimental): Participants will be given mobile- and hospital-based lifestyle interventions. The mobile-based interventions including dietary guidance, exercise supervision and weight monitoring will be conducted by trained physicians through WeChat group on cell phone every 1 to 2 weeks. Participants need to report their physical activity and weight information every week through WeChat group. Hospital-based intervention is a ≥5 minutes one-to-one and face-to-face personalized lifestyle counselling leading by a trained physician every 4 weeks during <14 weeks of gestation, every 2 weeks during 14-28 weeks of gestation, and once a week during ≥28 weeks of gestation. Participants' dietary information will be collected for any 3 consecutive days chosen by participants during 12-14 weeks of gestation, 24-28 weeks of gestation and >36 weeks of gestation respectively using a food frequency questionnaire.
  Interventions: Behavioral: mobile-based combining with hospital-based lifestyle interventions
- control group (No Intervention): Participants in control group will be managed in accordance with the standard practice.

INTERVENTIONS:
Behavioral: mobile-based combining with hospital-based lifestyle interventions — The same as that stated in arm descriptions.
  Arms: Lifestyle intervention group

SUMMARY:
This is a single-blind randomized controlled trial, aiming to evaluate the preventive effects of mobile-based combining with hospital-based lifestyle interventions on GDM among women with advanced maternal age. It will be conducted in Beijing, with a sample size of 346. All eligible pregnant women will be randomly assigned to either the intervention or control group, and followed up to delivery.

DETAILED DESCRIPTION:
After the adjustment of fertility policy in China, the prevalence of advanced maternal age (AMA) has become a crucial issue in maternal health care. AMA can greatly increase the risk of gestational diabetes mellitus (GDM) during pregnancy. However, there is still a lack of high-quality evidence on GDM preventive interventions for AMA pregnancy in China.

In this randomized study, the investigators aim to examine whether mobile-based combining with hospital-based lifestyle interventions have preventive effects on GDM in AMA pregnancies. The investigators will enroll a total of 346 singleton pregnant women in Peking University First Hospital and randomly assign them to either the intervention or control group. Information of maternal characteristics will be obtained at recruitment. At each prenatal visit, weight and blood pressure of all participants will be measured. For each participant, fasting venous blood samples will be collected at <14 weeks of gestation, 24-28 weeks of gestation and pre-labor, and respectively assayed for fasting plasma glucose, glycated hemoglobin. The primary outcome is the incidence of GDM. The secondary outcomes include maternal glycated hemoglobin level, maternal fasting plasma glucose level, maternal complications, pregnancy outcomes, etc.

ELIGIBILITY:
Inclusion Criteria:

* local resident in Beijing
* Singleton pregnancy
* Aged ≥35 years
* Overweight or obesity (Body mass index is between 24 and 27.9 kg/m2 or ≥28 kg/m2)
* ≤12 weeks of gestation
* written informed consent is obtained

Exclusion Criteria:

* Diagnosed with type 1 or type 2 diabetes before pregnancy
* Diagnosed with GDM or impaired glucose tolerance at enrollment
* use of medication that influences glucose metabolism currently, such as metformin, etc.
* multiple pregnancy
* current substance abuse
* unable to exercise due to physical disability
* diagnosed severe psychiatric disorder
* Other conditions not suitable for intervention as judged by physicians

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of gestational diabetes mellitus | from 24 weeks of gestation to delivery.
  diagnosed by the oral glucose tolerance test

SECONDARY OUTCOMES:
maternal glycated hemoglobin level | at <14 weeks of gestation, 24-28 weeks of gestation, and pre-labor
  obtained from fasting venous blood samples
maternal fasting plasma glucose level | at <14 weeks of gestation, 24-28 weeks of gestation, and pre-labor
  obtained from fasting venous blood samples
maternal gestational weight gain | from recruitment to delivery
  in kilograms
incidence of gestational hypertension | from 20 weeks of gestation to delivery.
  defined as a systolic blood pressure of ≥140 mmHg or diastolic blood pressure of ≥90 mmHg occurring after 20 weeks of gestation
incidence of pre-eclampsia | from 20 weeks of gestation to delivery.
  defined as a systolic blood pressure of ≥140 mmHg or diastolic blood pressure of ≥90 mmHg occurring after 20 weeks of gestation in a previously normotensive woman combined with new-onset proteinuria of ≥0.3 g/24 h
delivery mode | at delivery
  such as vaginal delivery, ceseran delivery, operative vaginal delivery
birthweight | at delivery
  in original scale (g) or z-score
Macrosomia | at delivery
  defined as a birth weight of > 4000 g
low birthweight | at delivery
  defined as a birth weight of < 2500 g
Gestational age at birth | at delivery
  in weeks
Premature delivery | at delivery
  less than 37 weeks' gestational age
Apgar score | 1 min and 5 min
  Apagr score
maternal dietary information | any 3 consecutive days chosen randomly by participants during 12-14 weeks of gestation, 24~28 weeks of gestation and >36 weeks of gestation respectively
  food species and servings
maternal physical activity information | every 1-2 weeks during enrollment to delivery
  type of physical activity and time spend on it weekly

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Wei, PhD, Principal Investigator — Peking University First Hospital; Yubo Zhou, Principal Investigator — Peking University
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared upon the request of other researchers, and all the key variables that will be reported in the main paper are planned to be shared
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After the publication of the main paper (hopefully before the end of 2024), the data will be available to share to other researchers
Access Criteria: Researchers should request the data via the following Email:
  zhouyubo@bjmu.edu.cn or weiyumei1982@126.com